CLINICAL TRIAL: NCT05686551
Title: A Phase II, Randomized, Double-blind, Placebo-controlled, Dose-finding Study to Evaluate the Safety, Biomarkers, and Efficacy of Tominersen in Individuals With Prodromal and Early Manifest Huntington's Disease
Brief Title: GENERATION HD2. A Study to Evaluate the Safety, Biomarkers, and Efficacy of Tominersen Compared With Placebo in Participants With Prodromal and Early Manifest Huntington's Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BN42489; Other (Other: GENERATION HD2); 2022-001991-32 (EudraCT Number); 2023-503928-10-00 (EU CTIS Number)
Record Dates: First submitted 2022-12-16; First posted 2023-01-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Huntington Disease
Keywords: Prodromal and Early Manifest Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — tominersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tominersen 60 milligrams (mg) (Experimental)
  Interventions: Drug: Tominersen 60 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Tominersen 100 mg (Experimental)
  Interventions: Drug: Tominersen 100 mg

INTERVENTIONS:
Drug: Tominersen 60 mg — 60 mg tominersen administered intrathecally every 16 weeks (Q16W).
  Other Names: RO7234292;; RG6042
  Arms: Tominersen 60 milligrams (mg)
Drug: Placebo — Matching placebo administered intrathecally Q16W.
  Arms: Placebo
Drug: Tominersen 100 mg — 100 mg tominersen administered intrathecally Q16W.
  Other Names: RO7234292;; RG6042
  Arms: Tominersen 100 mg

SUMMARY:
This study will evaluate the safety, biomarkers, and efficacy of tominersen compared with placebo in participants with prodromal and early manifest Huntington's Disease (HD).

ELIGIBILITY:
Inclusion Criteria

-HD gene expansion mutation carrier status with a cytosine-adenine-guanine-age product (CAP) score of 400-500 inclusive

Either:

* Prodromal HD (defined as Diagnostic Confidence Level (DCL) 2 to 3, Independence Scale (IS) ⩾70, and TFC ⩾8); or
* Early manifest HD (defined as DCL 4, IS ⩾70, and TFC ⩾8);
* Total body weight > 40 kilograms (kg) and a body mass index (BMI) within the range of 18-32 kilograms per meter square (kg/m2)
* Study companion

Exclusion Criteria

* Current or previous use of an antisense oligonucleotide (ASO) (including small interfering ribonucleic acid [RNA]) or any huntingtin gene/protein (HTT) lowering therapy (including tominersen)
* Anti-platelet or anticoagulant therapy within 14 days prior to screening or anticipated use during the study, including, but not limited to, aspirin (unless ≤ 81 milligrams per day [mg/day]), clopidogrel, dipyridamole, warfarin, dabigatran, rivaroxaban, apixaban, and heparin
* History of gene therapy, cell transplantation, or brain surgery
* Hydrocephalus
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 5 months after the final dose of study drug
* History of attempted suicide or suicidal ideation with plan (i.e., active suicidal ideation) that required hospital visit and/or change in level of care within 12 months prior to screening

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 301 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events (AEs), With Severity Determined According to the AE Severity Grading Scale | Up to approximately 24 months
Change From Baseline in Clinical Laboratory Results - Cerebrospinal Fluid (CSF) White Blood Cell (WBC) | From baseline visit (Day 1), and months 4, 8, 9, 12, 16
Change From Baseline in Clinical Laboratory Results CSF Protein | From baseline visit (Day 1), and months 4, 8, 9, 12, 16
Change From Baseline in Structural Magnetic Resonance Imaging (MRI) Assessing Any New Abnormalities Including Radiographic Features Consistent With Hydrocephalus and Other Relevant MRI Safety Findings | From baseline, months 4, 8, 12, 16 and up to approximately month 24
Percentage Change From Baseline in Geometric Means of CSF Mutant Huntingtin (mHTT) Protein Levels at Month 9 | Baseline, Month 9
Change From Baseline in Composite Unified Huntington's Disease Rating Scale (cUHDRS) Scores (non-U.S. Sites) at 16 Months | Baseline to 16 months
  Change in scores on the scale.
Change From Baseline in Total Functional Capacity (TFC) Scores (U.S. Sites) at 16 Months | Baseline to 16 months
  Change in scores on the scale.

SECONDARY OUTCOMES:
Change From Baseline in Montreal Cognitive Assessment (MoCA) Scores | From baseline, months 4, 8, 12, 16 and up to approximately month 24
Percentage of Participants With Suicidal Ideation or Behavior (I/B) as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) at Each Visit, Including Detailed Focus on Any Individual Cases Identified as Having Severe I/B During the Study Conduct | Up to approximately 24 months
Change From Baseline at 16 Months for the Assessments of TFC (non-U.S. Sites) Scores | Baseline to 16 months
Change From Baseline at 16 Months for the Assessments of cUHDRS (U.S. Sites) Scores | Baseline to 16 months
Change From Baseline at 16 Months for the Assessments of Symbol Digit Modalities Test (SDMT) Scores | Baseline to 16 months
Change From Baseline at 16 Months for the Assessments of Stroop Word Reading (SWR) Score | Baseline to 16 months
Change From Baseline at 16 Months for the Assessment of Total Motor Score (TMS) | Baseline to 16 months
Change From Baseline in CSF Neurofilament Light Chain (NfL) Levels at 16 Months | Baseline to 16 months
Incidence of Anti-drug Antibodies (ADAs) at Specified Timepoints Relative to the Prevalence of ADAs at Baseline | From baseline, months 4, 8, 12, 16 and up to approximately month 24
Titers Determined if ADAs are Identified | From baseline, months 4, 8, 12, 16 and up to approximately month 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (70):
- United States (18):
  - Uab Medicine, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California Davis Medical System, Sacramento, California
  - CenExel Rocky Mountain Clinical Research, LLC, Englewood, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Dent Neurological Institute, Amherst, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - EvergreenHealth Investigational Drug Services, Kirkland, Washington
  - Inland Northwest Research, Spokane, Washington
- Argentina (4):
  - CINME, Buenos Aires
  - Hospital Ramos Mejía, CABA
  - INEBA, Capital Federal
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
- Australia (3):
  - Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Perron Institute for Neurological and Translational Science, Nedlands, Western Australia
- Uniklinik fuer Neurologie, Medizinische Universitaet Innsbruck, Innsbruck, Austria
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Montreal Neurological Inst, Montreal, Quebec
- Rigshospitalet, Hukommelsesklinikken, København Ø, Denmark
- France (8):
  - CHU Angers, Batiement Larrey 2, Neurologie, Angers
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Hopital Henri Mondor, Créteil
  - Hopital Roger Salengro Service de Neurologie, Lille
  - CHU de la Timone - Hopital d Adultes, Marseille
  - Hopital Gui de Chauliac, Montpellier
  - CHU Strasbourg Hpital Hautepierre, Strasbourg
  - CHU toulouse - Hôpital Purpan, Toulouse
- Germany (8):
  - Uniklinik RWTH Aachen, Aachen
  - Charité - Universitätsmed. Berlin, Klinik für Psychiatrie und Psychotherapie, Berlin
  - St. Josef-Hospital, Neurologische Klinik der Ruhr-Uni, Bochum
  - German Center for Neurodegenerative Diseases (DZNE), Bonn
  - Universitätsklinikum Erlangen, Abteilung Molekulare Neurologie, Erlangen
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck, Lübeck
  - kbo - Isar-Amper-Klinikum Taufkirchen, Taufkirchen
  - Universitätsklinikum Ulm, Ulm
- Italy (3):
  - Ospedale Bellaria, Bologna, Emilia-Romagna
  - Azienda Ospedaliera Sant'Andrea, Rome, Lazio
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Lombardy
- New Zealand (2):
  - New Zealand Brain Research Institute, Christchurch
  - Waikato Hospital, Hamilton
- Poland (3):
  - Szpital Sw. Wojciecha, Gdansk
  - Krakowska Akademia Neurologii Sp z o.o. Centrum Neurologii K, Krakow
  - Wojskowy Instytut Medycyny Lotniczej, Warsaw
- Portugal (2):
  - Hospital de Santa Maria, Lisbon
  - CNS - Campus Neurológico, Torres Vedras
- Spain (7):
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Burgos. Servicio de Neurología, Burgos
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario la Fe, Valencia
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - Neurozentrum Siloah, Gümligen
- United Kingdom (6):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Addenbrookes Hospital, Cambridge
  - Chapel Allerton Hospital, Leeds
  - UCL Hospital NHS Trust, London
  - John Radcliffe Hospital, Oxford
  - Southampton University Hospitals NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing
Supporting Information: Study Protocol

REFERENCES:
- [Derived] McColgan P, Thobhani A, Boak L, Schobel SA, Nicotra A, Palermo G, Trundell D, Zhou J, Schlegel V, Sanwald Ducray P, Hawellek DJ, Dorn J, Simillion C, Lindemann M, Wheelock V, Durr A, Anderson KE, Long JD, Wild EJ, Landwehrmeyer GB, Leavitt BR, Tabrizi SJ, Doody R; GENERATION HD1 Investigators. Tominersen in Adults with Manifest Huntington's Disease. N Engl J Med. 2023 Dec 7;389(23):2203-2205. doi: 10.1056/NEJMc2300400. No abstract available. PMID 38055260